CLINICAL TRIAL: NCT05028101
Title: The Impact of Functional Medicine On Wound Healing From Delayed Autologous Breast Reconstruction - A Feasibility Study
Brief Title: The Impact of Functional Medicine On Wound Healing From Delayed Autologous Breast Reconstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4119
Record Dates: First submitted 2021-06-28; First posted 2021-08-31 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Standard of Care (SOC)) (Active Comparator): Reconstructive surgical technique, delayed autologous breast reconstruction, and usual local anesthesia and analgesia during hospital stay.
  Interventions: Procedure: Delayed autologous breast reconstruction
- SOC + Functional Medicine (Experimental): Reconstructive surgical technique, delayed autologous breast reconstruction, and usual local anesthesia and analgesia during hospital stay.
  Perioperative nutrition and lifestyle-based interventions along with select dietary supplements.
  Interventions: Procedure: Delayed autologous breast reconstruction; Behavioral: Perioperative Functional Medicine (FM) Care

INTERVENTIONS:
Procedure: Delayed autologous breast reconstruction — SOC: Delayed autologous breast reconstruction
Behavioral: Perioperative Functional Medicine (FM) Care — SOC plus FM: A food plan that encourages consumption of nutrient-dense whole foods. It provides adequate protein, balanced quality fats and foods which contain targeted nutrients essential to proper wound healing. Select dietary supplements will be provided as an adjunct to the food plan. Health coaching will support optimal sleep, adequate movement/exercise and stress reduction.
  Arms: SOC + Functional Medicine

SUMMARY:
This study will examine if a functional medicine approach, delivered as an adjunct to standard of care, is feasible, safe, clinically beneficial and cost-effective for patients undergoing autologous breast reconstruction.

DETAILED DESCRIPTION:
Autologous microsurgical breast reconstruction is associated with a protracted recovery and a significant amount of opioid utilization. Many institutions have "Enhanced Recovery After Surgery (ERAS)" protocols that utilize multi-modality therapy to decrease opioid use, length of stay, hospital costs and expedite recovery. However, nutrition-based interventions used perioperatively are not currently part of ERAS protocols for surgical sub-specialties, including breast surgery despite ample literature that nutrition (with or without supplements) can improve surgical wound healing and other outcomes.

The functional medicine model of care expands upon the conventional medicine model of care by providing a unique operating system that works to reverse illness, promote health and optimize function. A foundation of functional medicine is the use of food as medicine to prevent, treat and reverse chronic disease. Dietary supplements are used as an adjunct to nutrition-based interventions. Dietitians support patients with implementing food plans, and health coaches support patients through lifestyle and behavioral changes focused on sleep, exercise and movement and stress reduction.

This study will examine the feasibility of implementing a functional medicine-based intervention focused on nutrition and lifestyle, and the ability of the intervention to improve wound healing and decrease various post-operative complications in patients undergoing autologous breast reconstruction.

All participants will be asked to attend study visits, complete questionnaires and have their blood drawn. Participants randomized to standard of care plus functional medicine will be asked to also follow a specific food plan, take specific dietary supplements, exercise and engage in stress reduction techniques for 3 months prior to and after surgery. The study duration is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing uni- or bilateral delayed abdominally-based breast reconstruction at the Cleveland Clinic.
* Women of childbearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization) for the duration of the study.
* Capable of providing written informed consent prior to any protocol-specified procedures.
* Willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* BMI > 37
* Women who are pregnant, nursing, or planning pregnancy during the trial.
* Have a serious concomitant illness that could interfere with the subject's participation in the trial (allergy preventing supplement usage)
* Undergoing chemotherapy during proposed nutritional intervention (3 months before or after surgery).
* Are unable to or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access.
* Clinical diagnosis of cognitive impairment or dementia.
* Known sensitivity to nutritional supplements.
* History of being seen or had intervention/care in Functional Medicine or following Functional Medicine principles.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Feasibility defined by percent randomized. | Baseline
  Success will be defined as enrolling and randomizing 25% or more of those screened per arm.
Number of in-person visits completed. | Up to 26 weeks
  Number of in-person visits completed.
Number of virtual visits completed. | Up to 26 weeks
  Number of virtual visits completed.
Adherence to recommended dietary intervention. | Up to 26 weeks
  Percent of participants adhering to recommended dietary intervention.
Adherence to recommended lifestyle interventions. | Up to 26 weeks
  Percent of participants adhering to lifestyle interventions.
Adherence to prescribed dietary supplementation. | Up to 26 weeks
  Percent of participants adhering to prescribed dietary supplementation.
Percent completion of study-specific surveys. | Up to 26 weeks
  Percent of the following surveys completed:
  * BreastQ (baseline, wks 12, and 26)
  * PROMIS Questionnaire (baseline and wks 5, 12 and 26)
  * Medical Symptom Questionnaire (MSQ) (baseline and wks 5, 12 and 26)
  * Nutrition and Lifestyle Adherence Survey (randomization and then weekly for the duration of the study)
  * Dietary Supplementation Adherence Survey (only those randomized to SOC plus functional medicine; wk1 and then weekly for the duration of the study)
  Note: the BRA and SKIN surveys are not completed by the patient, but by the provider.
Number of Serious Adverse Events (SAE's). | Up to 26 weeks
  Number of Serious Adverse Events (SAE's).

SECONDARY OUTCOMES:
Number of re-operations for wound management. | Up to 26 weeks
  Number of re-operations for wound management (mean & standard deviation).
Number of hospital re-admissions. | Up to 26 weeks
  Number of hospital re-admissions (mean & standard deviation).
Length-of-stay upon hospital re-admission. | Up to 26 weeks
  Length-of-stay upon hospital re-admission (mean & standard deviation).
Number of antibiotic prescriptions. | Up to 26 weeks
  Infection rates assessed by number of antibiotic prescriptions (mean & standard deviation). Standard of care (SOC), post-surgery prophylactic antibiotic prescriptions will not be considered.
Correlate all post-operative complications with the predicted risk from the BRA scoring system. | Up to 26 weeks
  Surgical complications will be measured within each arm and the predicted risk will be compared to the actual incidence. Surgical complications is defined as the total number of all the complications (eg. surgical site infection, seroma, dehiscence, flap loss and reoperation). The minimum and maximum probabilities of experiencing surgical complications based on the BRA scoring system are 11.7% and 57.9%, respectively. The American Society of Plastic Surgeons Tracking Operations and Outcomes for Plastic Surgeons (TOPS) database which tracks 30-day outcomes for plastic surgery was used to determine the minimum and maximum probabilities of this complication.
Correlate post-operative surgical site infection complications with the predicted risk from the BRA scoring system. | Up to 26 weeks
  Surgical site infection (SSI) will be measured within each arm and the predicted risk will be compared to the actual incidence. SSI is defined as a superficial SSI or deep incisional SSI.
  The minimum and maximum probabilities of experiencing a SSI based on the BRA scoring system are 2.7% and 54.8%, respectively. The American College of Surgeons National Surgical Quality Improvement Program (NSQIP) database which tracks 30-day outcomes for plastic surgery was used to determine the minimum and maximum probabilities of this complication.
Correlate post-operative seroma complications with the predicted risk from the BRA scoring system. | Up to 26 weeks
  Seroma will be measured within each arm and the predicted risk will be compared to the actual incidence. Seroma is defined as a fluid collection that develops after surgery necessitating aspiration or surgical intervention. The minimum and maximum probabilities of experiencing a seroma based on the BRA scoring system are 1.8% and 13.8%, respectively. The American Society of Plastic Surgeons Tracking Operations and Outcomes for Plastic Surgeons (TOPS) database which tracks 30-day outcomes for plastic surgery was used to determine the minimum and maximum probabilities of this complication.
Correlate post-operative dehiscence complications with the predicted risk from the BRA scoring system. | Up to 26 weeks
  Dehiscence will be measured within each arm and the predicted risk will be compared to the actual incidence. Dehiscence is defined as separation of the layers of a surgical wound, which may be partial or complete with disruption of the fascia. The minimum and maximum probabilities of experiencing dehiscence based on the BRA scoring system are 3.7% and 50.2%, respectively. The American Society of Plastic Surgeons Tracking Operations and Outcomes for Plastic Surgeons (TOPS) database which tracks 30-day outcomes for plastic surgery was used to determine the minimum and maximum probabilities of this complication.
Correlate post-operative flap loss complications with the predicted risk from the BRA scoring system. | Up to 26 weeks
  Flap loss will be measured within each arm and the predicted risk will be compared to the actual incidence. Flap loss is defined as complete removal of flap after complication. The minimum and maximum probabilities of experiencing flap loss based on the BRA scoring system are 4.3% and 49.6%, respectively. The American Society of Plastic Surgeons Tracking Operations and Outcomes for Plastic Surgeons (TOPS) database which tracks 30-day outcomes for plastic surgery was used to determine the minimum and maximum probabilities of this complication.
Correlate post-operative reoperation complications with the predicted risk from the BRA scoring system. | Up to 26 weeks
  Reoperation will be measured within each arm and the predicted risk will be compared to the actual incidence. Reoperation is defined as a return to operating room for a procedure. This does not refer to procedures performed in the office under local. The minimum and maximum probabilities of experiencing reoperation based on the BRA scoring system are 4.3% and 23.0%, respectively. The American Society of Plastic Surgeons Tracking Operations and Outcomes for Plastic Surgeons (TOPS) database which tracks 30-day outcomes for plastic surgery was used to determine the minimum and maximum probabilities of this complication.
Evaluate narcotic utilization while in the hospital. | While in hospital, an average of 3 days
  Morphine utilization (Oral morphine equivalents (mg)).
Evaluate narcotic utilization while in the hospital. | While in hospital, an average of 3 days
  Morphine utilization (Oral morphine equivalents (mg/kg)).
Evaluate narcotic utilization while in the hospital. | While in hospital, an average of 3 days
  Morphine utilization (Oral morphine equivalents (mg/kg/day)).
Evaluate narcotic utilization while in the hospital. | While in hospital, an average of 3 days
  Morphine utilization (IV morphine equivalents (mg)).
Evaluate narcotic utilization while in the hospital. | While in hospital, an average of 3 days
  Morphine utilization (IV morphine equivalents (mg/kg)).
Evaluate narcotic utilization while in the hospital. | While in hospital, an average of 3 days
  Morphine utilization (IV morphine equivalents (mg/kg/day).
Evaluate narcotic utilization while in the hospital. | While in hospital, an average of 3 days
  Morphine utilization (total morphine equivalents (mg) while in hospital.
Evaluate narcotic utilization while in the hospital. | While in hospital, an average of 3 days
  Morphine utilization (total morphine equivalents (mg/kg) while in hospital.
Evaluate narcotic utilization while in the hospital. | While in hospital, an average of 3 days
  Morphine utilization (total morphine equivalents (mg/kg/day) while in hospital.
Change in Complete Blood Count with Differential (CBC). | Baseline to 12 weeks
  Change in CBC (mean & standard deviation).
Change in Complete Blood Count with Differential (CBC). | Baseline to 26 weeks
  Change in CBC (mean & standard deviation).
Change in Comprehensive Metabolic Pane (CMP). | Baseline to 12 weeks
  Change in CMP (mean & standard deviation).
Change in Comprehensive Metabolic Pane (CMP). | Baseline to 26 weeks
  Change in CMP (mean & standard deviation).
Change in Hemoglobin A1c (HbA1c). | Baseline to 12 weeks
  Change in % HbA1c (mean & standard deviation).
Change in Hemoglobin A1c (HbA1c). | Baseline to 26 weeks
  Change in % HbA1c (mean & standard deviation).
Change in nuclear magnetic resonance (NMR) LipoProfile. | Baseline to 12 weeks
  Change in NMR LipoProfile (mean & standard deviation).
  LDL Particle Number (L): (Normal Range: < 1000 nmol) LDL Cholesterol (dL): (Normal Range: 0 - 99 mg) HDL Cholesterol (dL) : (Normal Range: >39 mg) Triglycerides (dL): (Normal Range: 0 - 149 mg) Total Cholesterol (dL): (Normal Range: 100 - 199 mg) Total HDL Particles (L): (Normal Range: >=30.5 umol) Small LDL-P (L): (Normal Range: < =527 nmol) Large VLDL-P (L): (Normal Range: < =2.7 nmol/L) Large HDL-P (L): (Normal Range: >=4.8 umol) VLDL Size (nm): (Normal Range: < =46.6 nm) LDL Size (nm): (Normal Range: >20.5 nm) HDL Size (nm): (Normal Range: >=9.2 nm) LP/IR Score: (Normal Range: < =45)
Change in NMR LipoProfile. | Baseline to 26 weeks
  Change in NMR LipoProfile (mean & standard deviation).
  LDL Particle Number (L): (Normal Range: < 1000 nmol) LDL Cholesterol (dL): (Normal Range: 0 - 99 mg) HDL Cholesterol (dL) : (Normal Range: >39 mg) Triglycerides (dL): (Normal Range: 0 - 149 mg) Total Cholesterol (dL): (Normal Range: 100 - 199 mg) Total HDL Particles (L): (Normal Range: >=30.5 umol) Small LDL-P (L): (Normal Range: < =527 nmol) Large VLDL-P (L): (Normal Range: < =2.7 nmol/L) Large HDL-P (L): (Normal Range: >=4.8 umol) VLDL Size (nm): (Normal Range: < =46.6 nm) LDL Size (nm): (Normal Range: >20.5 nm) HDL Size (nm): (Normal Range: >=9.2 nm) LP/IR Score: (Normal Range: < =45)
Change in high-sensitivity C-Reactive Protein (hsCRP). | Baseline to 12 weeks
  Change in hsCRP (mean & standard deviation).
Change in high-sensitivity C-Reactive Protein (hsCRP). | Baseline to 26 weeks
  Change in hsCRP (mean & standard deviation).
Change in Vitamin D. | Baseline to 12 weeks
  Change in Vitamin D (ng/mL) (mean & standard deviation).
Change in Vitamin D. | Baseline to 26 weeks
  Change in Vitamin D (ng/mL) (mean & standard deviation).
Change in OmegaCheck. | Baseline to 12 weeks
  Change in OmegaCheck (mean & standard deviation).
  Arachidonic Acid (% by wt) Arachidonic Acid/EPA ratio Docosahexaenoic acid (DHA) (% by wt) Docosapentaenoic acid (DPA) (% by wt) Eicosapentaenoic acid (EPA) (% by wt) Linoleic Acid (% by wt) Omega-3 total (% by wt) Omega-6 total (% by wt) Omega-6/3 Ratio OmegaCheck (total EPA+DPA+DHA reported as % by wt)
Change in OmegaCheck. | Baseline to 26 weeks
  Change in OmegaCheck (mean & standard deviation).
  Arachidonic Acid (% by wt) Arachidonic Acid/EPA ratio Docosahexaenoic acid (DHA) (% by wt) Docosapentaenoic acid (DPA) (% by wt) Eicosapentaenoic acid (EPA) (% by wt) Linoleic Acid (% by wt) Omega-3 total (% by wt) Omega-6 total (% by wt) Omega-6/3 Ratio OmegaCheck (total EPA+DPA+DHA reported as % by wt)
Total healthcare costs. | At 26 weeks
  Measure cost of laboratory testing, dietary supplementation, initial hospital length of stay, and post-surgical complications requiring intervention (if applicable).
Net change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Physical Health (GPH) scores. | Baseline to week 12
  Change in PROMIS GPH scores (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes
Net change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Physical Health (GPH) scores. | Baseline to week 26
  Change in PROMIS GPH scores (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes
Net change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Physical Health (GPH) scores. | Baseline to week 5
  Change in PROMIS GPH scores (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
Clinically-meaningful change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Physical Health (GPH) scores. | Baseline to week 5
  Clinically-meaningful change in PROMIS GPH, or improvements in 5.00 points or more (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
  Improvement: ≥5.00 points Slightly Better: 2.50 to 4.99 points Similar: -2.49 to 2.49 points Slightly Worse: -2.50 to -4.99 points
Clinically-meaningful change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Physical Health (GPH) scores. | Baseline to week 12
  Clinically-meaningful change in PROMIS GPH, or improvements in 5.00 points or more (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
  Improvement: ≥5.00 points Slightly Better: 2.50 to 4.99 points Similar: -2.49 to 2.49 points Slightly Worse: -2.50 to -4.99 points
Clinically-meaningful change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Physical Health (GPH) scores. | Baseline to week 26
  Clinically-meaningful change in PROMIS GPH, or improvements in 5.00 points or more (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
  Improvement: ≥5.00 points Slightly Better: 2.50 to 4.99 points Similar: -2.49 to 2.49 points Slightly Worse: -2.50 to -4.99 points
Change in mean value of the continuous variable of PROMIS GPH. | Baseline to week 5
  Change in mean value of the continuous variable of PROMIS GPH.
Change in mean value of the continuous variable of PROMIS GPH. | Baseline to week 12
  Change in mean value of the continuous variable of PROMIS GPH.
Change in mean value of the continuous variable of PROMIS GPH. | Baseline to week 26
  Change in mean value of the continuous variable of PROMIS GPH.
Net change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Mental Health (GMH). | Baseline to week 5
  Change in PROMIS GMH scores (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
Net change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Mental Health (GMH). | Baseline to week 12
  Change in PROMIS GMH scores (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
Net change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Mental Health (GMH). | Baseline to week 26
  Change in PROMIS GMH scores (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
Clinically-meaningful change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Mental Health (GMH) scores. | Baseline to week 5
  Clinically-meaningful change in PROMIS GMH, or improvements in 5.00 points or more (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
  Improvement: ≥5.00 points Slightly Better: 2.50 to 4.99 points Similar: -2.49 to 2.49 points Slightly Worse: -2.50 to -4.99 points
Clinically-meaningful change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Mental Health (GMH) scores. | Baseline to week 12
  Clinically-meaningful change in PROMIS GMH, or improvements in 5.00 points or more (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
  Improvement: ≥5.00 points Slightly Better: 2.50 to 4.99 points Similar: -2.49 to 2.49 points Slightly Worse: -2.50 to -4.99 points
Clinically-meaningful change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Mental Health (GMH) scores. | Baseline to week 26
  Clinically-meaningful change in PROMIS GMH, or improvements in 5.00 points or more (mean & standard deviation).
  PROMIS is an NIH-validated set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children within the general population and in those living with chronic conditions. This is considered SOC for the Center for Functional Medicine. Scores are transformed into T-Scores. The mean (SD) of the US General Population is 50 (10). Higher scores mean better outcomes.
  Improvement: ≥5.00 points Slightly Better: 2.50 to 4.99 points Similar: -2.49 to 2.49 points Slightly Worse: -2.50 to -4.99 points
Change in mean value of the continuous variable of PROMIS GMH. | Baseline to week 5
  Change in mean value of the continuous variable of PROMIS GMH.
Change in mean value of the continuous variable of PROMIS GMH. | Baseline to week 12
  Change in mean value of the continuous variable of PROMIS GMH.
Change in mean value of the continuous variable of PROMIS GMH. | Baseline to week 26
  Change in mean value of the continuous variable of PROMIS GMH.
Change in Breast-Q scores. | Baseline to week 12
  Change in Breast-Q score (mean & standard deviation).
  Breast-Q is a validated comprehensive evaluation of breast health and wellness. Transformed scores range from 0-100 with higher score means greater satisfaction or better QoL.
Change in Breast-Q scores. | Baseline to week 26
  Change in Breast-Q score (mean & standard deviation).
  Breast-Q is a validated comprehensive evaluation of breast health and wellness. Transformed scores range from 0-100 with higher score means greater satisfaction or better QoL.
Change in Medical System Questionnaire (MSQ) scores. | Baseline to week 5
  Change participant's global symptoms measured by change in MSQ scores (mean & standard deviation).
  The MSQ identifies symptoms that a patient has experienced over the previous 48 hours based upon their health profile. The MSQ utilizes a semantic differential scale to determine how often a patient is experiencing a specific symptom and to track a participant's progress. All scores are totaled and higher MSQ scores indicate worsening of symptoms while lower scores indicate symptom improvement. This is considered SOC for the Center for Functional Medicine.
  Total Score Range: 0-352, with higher scores meaning worse outcomes.
Change in Medical System Questionnaire (MSQ) scores. | Baseline to week 12
  Change participant's global symptoms measured by change in MSQ scores (mean & standard deviation).
  The MSQ identifies symptoms that a patient has experienced over the previous 48 hours based upon their health profile. The MSQ utilizes a semantic differential scale to determine how often a patient is experiencing a specific symptom and to track a participant's progress. All scores are totaled and higher MSQ scores indicate worsening of symptoms while lower scores indicate symptom improvement. This is considered SOC for the Center for Functional Medicine.
  Total Score Range: 0-352, with higher scores meaning worse outcomes.
Change in Medical System Questionnaire (MSQ) scores. | Baseline to week 26
  Change participant's global symptoms measured by change in MSQ scores (mean & standard deviation).
  The MSQ identifies symptoms that a patient has experienced over the previous 48 hours based upon their health profile. The MSQ utilizes a semantic differential scale to determine how often a patient is experiencing a specific symptom and to track a participant's progress. All scores are totaled and higher MSQ scores indicate worsening of symptoms while lower scores indicate symptom improvement. This is considered SOC for the Center for Functional Medicine.
  Total Score Range: 0-352, with higher scores meaning worse outcomes.
Change in Nutrition and Lifestyle Adherence Survey scores. | Baseline to week 12
  Nutrition and lifestyle changes as measured by changes in Nutrition and Lifestyle Adherence Survey scores, which assesses participant diet, exercise and stress management in the prior week.
  Nutrition: Range of available points: 0-45 (higher = better) Sleep: Range of available points: 0-3 points (higher = better) Exercise/Movement: Range of available points: 0-20 points (higher = better) Stress Management: 0-8 points (higher = better) Total Composite Score Range: 0-76 (higher = better)
Change in Nutrition and Lifestyle Adherence Survey scores. | Baseline to week 26
  Nutrition and lifestyle changes as measured by changes in Nutrition and Lifestyle Adherence Survey scores, which assesses participant diet, exercise and stress management in the prior week.
  Nutrition: Range of available points: 0-45 (higher = better) Sleep: Range of available points: 0-3 points (higher = better) Exercise/Movement: Range of available points: 0-20 points (higher = better) Stress Management: 0-8 points (higher = better) Total Composite Score Range: 0-76 (higher = better)
Change in Dietary Supplement Adherence Survey scores. | Baseline to week 12
  Dietary supplementation use as part of the study measured by change Dietary Supplement Adherence Survey scores.
  O.N.E Omega: 0-4 points Probiotic 50B: 0-4 points Vitamin D3: 0-4 points Whey Basics: 0-4 points Curcumin with Bioperine: 0-4 points Zinc 30: 0-4 points Bromelain: 0-4 points
  * Only taken 1 week prior to and after surgery Total Score Range: 0-24 (except for the 1 week prior to and after surgery when the total score range is: 0-28, higher = better)
Change in Dietary Supplement Adherence Survey scores | Baseline to week 26
  Dietary supplementation use as part of the study measured by change Dietary Supplement Adherence Survey scores.
  O.N.E Omega: 0-4 points Probiotic 50B: 0-4 points Vitamin D3: 0-4 points Whey Basics: 0-4 points Curcumin with Bioperine: 0-4 points Zinc 30: 0-4 points Bromelain: 0-4 points
  * Only taken 1 week prior to and after surgery Total Score Range: 0-24 (except for the 1 week prior to and after surgery when the total score range is: 0-28 higher = better)
Number of days wounds necessitate dressing changes or packing post-surgery. | At 26 weeks
  Evaluation of wound healing by by assessing the number of days wounds necessitate dressing changes or packing post-surgery (mean & standard deviation).
SKIN Survey composite scores. | At 14 weeks
  The SKIN Survey composite score assesses severity and extent of mastectomy skin flap necrosis (MSFN) (eg. A1, B3, D2, etc.).
  Depth of MSFN is assessed from A to D:
  A = None, no evidence of MSFN B = Color change of skin flap suggesting impaired perfusion or ischemic injury (may be cyanosis or erythema) C = Partial thickness skin flap necrosis resulting in at least epidermal sloughing D = Full thickness skin flap necrosis
  Surface area of MSFN (%) is assessed by providing a value from 1 to 4:
  1. - None 0%
  2. - Breast, change affects 1-10% of breast skin or NAC, change affects 1-10% of nipple-areolar complex
  3. - Breast, change affects 11-30 % of breast skin or NAC, 11-30% of NAC affected, or total nipple involvement
  4. - Change affects >30% of breast skin or 30% of NAC
SKIN Survey composite scores. | At 15 weeks
  The SKIN Survey composite score assesses severity and extent of mastectomy skin flap necrosis (MSFN) (eg. A1, B3, D2, etc.).
  Depth of MSFN is assessed from A to D:
  A = None, no evidence of MSFN B = Color change of skin flap suggesting impaired perfusion or ischemic injury (may be cyanosis or erythema) C = Partial thickness skin flap necrosis resulting in at least epidermal sloughing D = Full thickness skin flap necrosis
  Surface area of MSFN (%) is assessed by providing a value from 1 to 4:
  1. - None 0%
  2. - Breast, change affects 1-10% of breast skin or NAC, change affects 1-10% of nipple-areolar complex
  3. - Breast, change affects 11-30 % of breast skin or NAC, 11-30% of NAC affected, or total nipple involvement
  4. - Change affects >30% of breast skin or 30% of NAC
SKIN Survey composite scores. | At 17 weeks
  The SKIN Survey composite score assesses severity and extent of mastectomy skin flap necrosis (MSFN) (eg. A1, B3, D2, etc.).
  Depth of MSFN is assessed from A to D:
  A = None, no evidence of MSFN B = Color change of skin flap suggesting impaired perfusion or ischemic injury (may be cyanosis or erythema) C = Partial thickness skin flap necrosis resulting in at least epidermal sloughing D = Full thickness skin flap necrosis
  Surface area of MSFN (%) is assessed by providing a value from 1 to 4:
  1. - None 0%
  2. - Breast, change affects 1-10% of breast skin or NAC, change affects 1-10% of nipple-areolar complex
  3. - Breast, change affects 11-30 % of breast skin or NAC, 11-30% of NAC affected, or total nipple involvement
  4. - Change affects >30% of breast skin or 30% of NAC
Average incision length. | At 14 weeks
  Wound healing as measured by average incision length (mean & standard deviation).
Average incision length. | At 15 weeks
  Wound healing as measured by average incision length (mean & standard deviation).
Average incision length. | At 17 weeks
  Wound healing as measured by average incision length (mean & standard deviation).
Average dehiscence length. | At 14 weeks
  Wound healing as measured by average dehiscence length (separation of the incision line) (mean & standard deviation).
Average dehiscence length. | At 15 weeks
  Wound healing as measured by average dehiscence (separation of the incision line) length (mean & standard deviation).
Average dehiscence length. | At 17 weeks
  Wound healing as measured by average dehiscence (separation of the incision line) length (mean & standard deviation).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Shallcross, ND, MPH, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share Individual Participant Data (IPD)